CLINICAL TRIAL: NCT02839642
Title: RIVA-PSP: Efficacy of Rivastigmine on Motor, Cognitive and Behavioural Impairment in Progressive Supranuclear Palsy: A Randomised Double Blind Placebo-controlled Clinical Trial
Brief Title: Efficacy of RIVAstigmine on Motor, Cognitive and Behavioural Impairment in Progressive Supranuclear Palsy
Acronym: RIVA-PSP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-11; 2016-001319-19 (EudraCT Number)
Record Dates: First submitted 2016-06-30; First posted 2016-07-21 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Progressive Supranuclear Palsy (PSP)
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivastigmine (Active Comparator): Subject will receive a treatment of Rivastigmine twice daily during 24 weeks of treatment.
  Study drug will be administered orally. Sufficient test drug will be dispensed to subjects or their caregivers at each study visit to allow twice daily dosing until the next scheduled study visit
  Interventions: Drug: Rivastigmine
- Placebo (Placebo Comparator): Subject will receive a placebo twice daily during 24 weeks of treatment. Study drug will be administered orally. Sufficient test drug will be dispensed to subjects or their caregivers at each study visit to allow twice daily dosing until the next scheduled study visit
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivastigmine
  Arms: Rivastigmine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Progressive supranuclear palsy (PSP) is a rare neurodegenerative disease from the parkinsonian syndrome group. It represents 5 to 10% of all parkinsonian syndromes and affects 3,000 to 10,000 persons in France. PSP is characterised by a doparesistant parkinsonism with axial signs such as early gait instability and falls, oculomotor signs such as a vertical gaze palsy, dysphagia and dysarthria, and both cognitive and behavioural disturbances. The latter predominantly manifest as psycho-motor slowness, apathy and frontal executive deficits. Swallowing impairments and falls may lead to life-threatening situations and death occurs 6-9 years after disease onset.

Apart from L-dopa which may transiently and inconsistently improve motor symptoms no effective symptomatic, disease-modifying or neuroprotective therapy is presently available to reduce disability in any way. Therefore these patients often receive mostly non-medical care such as physiotherapy and speech therapy.

In addition to dopaminergic degeneration there is evidence of cholinergic deficits in PSP correlated with gait and balance impairments . This stands in contrast with the limited number of studies of cholinergic augmentation strategies in PSP.

Trials of cholinesterase inhibitors in PSP have produced rather conflicting results: donepezil improves cognition but deteriorates some motor functions whereas a case series of 5 PSP patients treated with rivastigmine found an improvement in several cognitive aspects and no deterioration of motor functions .On the other hand in Parkinson's disease there is convincing evidence of a positive effect of rivastigmine on cognition , apathy and falls Investigators' hypothesis is that rivastigmine (an acetyl- and butyryl-cholinesterase inhibitor) may reduce gait and postural impairment in PSP and may therefore limit the number of falls and their consequences both in terms of injuries sustained (fractures etc...) and on the patients' autonomy. In addition investigators hypothesise that rivastigmine may also reduce the cognitive and behavioural impairment associated with PSP. Taken together these improvements are likely to produce a significant effect on the patients' quality of life and their caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* Probable PSP of the Richardson subtype as defined by the NINDS-SPSP criteria modified so as to allow inclusions of patients who have first fallen within 3 years of disease onset.
* Aged 41 to 80 years at the time of screening
* Judged by site investigator to be able to comply with gait/balance and neuropsychological evaluations at baseline and throughout the study
* Able to ambulate independently or with assistance (cane)
* Score ≥ 20 on the mini-mental state examination (MMSE) at screening
* A reliable caregiver - defined as a person having frequent contact with subject (≥ 3 hours per day) and willing to fill the fall diaries and monitor study medication compliance and the subject's health and concomitant medication throughout the study - must accompany the subject to all visits.
* A fall or near fall rate ≥ 2/week in average (estimated through interview at screening and confirmed during a 2-week period between screening and baseline using fall postcards).
* Any parkinsonian medication taken by the subject must be stable in dose for 4 weeks prior to screening and must remain stable for the duration of the study
* Stable on all other chronic medications for 4 weeks prior to screening
* Written informed consent provided by subject and caregiver.

Exclusion Criteria:

* Non ambulatory patient.
* History and clinical examination suggesting another parkinsonian syndrome (Parkinson's disease, Dementia with Lewy Bodies, Corticobasal Degeneration, Multisystem Atrophy, Vascular Parkinsonism, tumoral parkinsonism, anti-psychotic drug-induced parkinsonism)
* Presence of other significant neurological or psychiatric disorders: Alzheimer's disease, epilepsy, history of stroke, psychotic disorder, severe bipolar or unipolar disorder
* A fall or near fall rate < 2/week in average (during a 2-week period between screening and baseline using fall postcards).
* Insufficient fluency in local language to complete neuropsychological, global and gait/balance assessments
* Score < 20 on the mini-mental state examination at screening
* Within 4 weeks of screening or during the course of the study concurrent treatment with any cholinesterase inhibitor medication (donepezil, galantamine, rivastigmine) or any cholinergic agent (agonist or antagonist) including memantine.
* History of deep brain stimulation surgery.
* Within 4 weeks of screening or during the course of the study concurrent treatment with beta blockers, any antipsychotic drugs or mood stabilisers.
* Any malignancy within 5 years of screening or current significant - judged as such by the site investigator - hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal, or neurological disease.
* Presence of an active gastro-duodenal ulcer, unstable asthma or chronic obstructive pulmonary disease.
* History of or current urinary retention requiring either anticholinergic medication or urethral catheterisation.
* The systolic blood pressure measurement is > 190 or < 85 mm Hg and/or the diastolic blood pressure measurement is > 105 or < 50 mm Hg at screening.
* Clinically significant laboratory abnormalities at screening, including creatinine ≥ 2.5 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times the upper limit of the normal reference range.
* The ECG is abnormal at screening and judged to be clinically significant by the site investigator. Particular attention will be given to any sign suggesting conduction disorders.
* Treatment with any investigational drugs or device within 60 days of screening.
* Ongoing pregnancy or lactation. Women with childbearing potential not using any form of efficacious contraception.
* Any contraindication for rivastigmine as defined by the ANSM
* Known hypersensitivity to rivastigmine or any cholinesterase inhibitor medication.

Ages: 41 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed at 4 months as the change from baseline of the number of falls and near falls over the past 2 week | baseline, 2 weeks, 4 months
  Efficacy will be assessed at 4 months as the change from baseline of the number of falls and near falls over the past 2 weeks using fall postcards sent weekly and filled daily by the subject and caregiver. The number of falls and near-falls will be expressed both as the total number of occurrences over that period and as the number of occurrence adjusted to the distance and number of hours walked (assessed using continuous accelerometer recordings)

SECONDARY OUTCOMES:
Change from baseline at 4 months measured by the global ans sub scores of the PSPRS scale (Progressive Supranuclear Palsy Rating Scale) | Baseline and 4 months
Change from baseline at 4 months measured by the Clinical Global Impression scale (patient and caregiver) | Baseline and 4 months
Apathy assessed using the Lille Apathy Rating Scale (LARS) both subject and caregiver versions | Baseline and 4 months
Assessment of the Quality of life of patient using the PSP-Quality of Life Scale (PSP-QoL) | Baseline and 4 months
Assessment of the Quality of life of patient using the EQ-5D | Baseline and 4 months
Assessment of the Quality of life of the caregiver using the PSP-Quality of Life Scale (PSP-QoL) | Baseline and 4 months
Assessment of the Quality of life of the caregiver using the EQ-5D | Baseline and 4 months
Caregiver burden assessed using the Caregiver Reaction Assessement (CRA) | Baseline and 4 months
Safety: recording of adverse events at each study visit and at the phone calls | 4 months
  Vital signs, laboratory tests and ECGs will be performed at each study visit to monitor any biological or cardiac adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service de Neurologie et Pathologie du Mouvement Hôpital de La Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided